CLINICAL TRIAL: NCT04214171
Title: Kinematics and Muscle Strength in Two, Five or 10 Years Afther Total Hip Arthroplasty: Comparison With Healthy Individuales Controlled Cross Sectional Study
Brief Title: Kinematics and Muscle Strength in Two, Five or 10 Years Afther Total Hip Arthroplasty
Acronym: Arthroplasty
Status: Completed | Type: Observational
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Vera Lucia dos Santos Alves, Head of Physical Therapy and Professor, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Other Study IDs: Joao B
Record Dates: First submitted 2018-01-03; First posted 2020-01-02 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Gait

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group 2 years: The group underwent total hip arthroplasty at 2 years
  Interventions: Diagnostic Test: Gait and muscle strength will be assessed
- group 5 years: The group underwent total hip arthroplasty at 5 years
  Interventions: Diagnostic Test: Gait and muscle strength will be assessed
- group 10 years: The group underwent total hip arthroplasty at 10 years
  Interventions: Diagnostic Test: Gait and muscle strength will be assessed
- group control: healthy patients
  Interventions: Diagnostic Test: Gait and muscle strength will be assessed

INTERVENTIONS:
Diagnostic Test: Gait and muscle strength will be assessed — The extensor moment of the hip during gait and evaluation of the muscular strength of the hip will be evaluated

SUMMARY:
Introduction: Femoral and acetabular replacement is characterized as total hip arthroplasty (THA). It has been used as treatment of various pathologies of this joint. In the postoperative period, some studies have shown that strength, function, range of motion and lower limb mechanics remains altered for more than One year after THA in relation to the non-operated side. However, studies that have correlated kinematics and hip muscle strength in individuals who underwent THA for long time, do not exist in literature. Objective: to evaluate lower limb muscle strength and 2D kinematics during stair ascending and descending in patients undergoing total hip arthroplasty. Methods: Third individuals who underwent total hip arthroplasty (THA) will be recruited at two, five and 10 year postoperative periods. They were allocated in three groups: Group 1 (10n), subjects submitted to THA for two years, Group 2 (10n) subjects submitted to THA for five years, Group 3 (10n) subjects submitted to THA for 10 years and Group 4 (10n) subjects without orthopaedic afections, all will be evaluated for dynamometric isometric muscle strength and kinematic analysis of stair ascending and descending by a "blinded" physical Therapist.

ELIGIBILITY:
Inclusion Criteria:

* The investigators will recruit 40 individuals who underwent total hip arthroplasty (THA) by the hospital hip surgery group in the periods of two, five and 10 years postoperatively
* Control group without orthopaedic afections. Inclusion criteria: patients submitted to total hip arthroplasty between two years (24 months - 35 months), five years (60 months - 71 months) and 10 years (120 months - 131 months), aged between 50 and 80 years and sign the terms of free and informed consent

Exclusion Criteria:

* patients with a history of prosthesis dislocations or revision of arthroplasty
* hip or lower limb pain
* asymmetry of the lower limbs greater than two centimeters
* previous surgeries in the lower limbs
* limited range of motion in the hip joint
* use of antidepressive drugs or analgesics for continuous use
* Presence of neuromuscular pathologies and functional incapacity to perform the activities proposed in the Kinematics analysis.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 individuals who underwent total hip arthroplasty (THA) by the hospital hip surgery group
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
kinematic analysis of hip movements for flexion | evaluated at 10 years after hip arthroplasty
  Analysis of the movements of the hip - range of motion for flexion
kinematic analysis of hip movements for extension | evaluated at 10 years after hip arthroplasty
  Analysis of the movements of the hip - range of motion for extension
kinematic analysis of hip movements for internal rotation | evaluated at 10 years after hip arthroplasty
  Analysis of the movements of the hip - range of motion for internal rotation
kinematic analysis of hip movements external rotation | evaluated at 10 years after hip arthroplasty
  Analysis of the movements of the hip - range of motion for external rotation

CONTACTS AND LOCATIONS:
Overall Officials: Vera Lucia Santos Alves, Dr, Study Director — Faculdade de Ciências Médicas da Santa Casa de São Paulo
Locations (1):
- João Barboza, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Foucher KC, Cinnamon CC, Ryan CA, Chmell SJ, Dapiton K. Hip abductor strength and fatigue are associated with activity levels more than 1 year after total hip replacement. J Orthop Res. 2018 May;36(5):1519-1525. doi: 10.1002/jor.23783. Epub 2017 Nov 28. PMID 29077218